CLINICAL TRIAL: NCT02861404
Title: Evaluation of Viral Status of Patients With Plantar Warts Included in VRAIE Study, Non-responder to Study Treatment
Acronym: BIOVRAIE
Status: Terminated | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: BIOVRAIE
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Plantar Warts
Keywords: HPV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Salicylate ointment: patients included in VRAIE study, treated with salicylate ointment (VRAIE study, NCT01059110)
  Interventions: Genetic: skin flakes collection
- Imiquimod: patients included in VRAIE study, treated with Imiquimod (VRAIE study, NCT01059110)
  Interventions: Genetic: skin flakes collection
- 5-Fluoro-Uracil: patients included in VRAIE study, treated with 5-Fluoro-Uracil (VRAIE study, NCT01059110)
  Interventions: Genetic: skin flakes collection
- Cryotherapy: patients included in VRAIE study, treated with cryotherapy (VRAIE study, NCT01059110)
  Interventions: Genetic: skin flakes collection
- placebo: patients included in VRAIE study, receiving placebo (VRAIE study, NCT01059110)
  Interventions: Genetic: skin flakes collection

INTERVENTIONS:
Genetic: skin flakes collection — viral status assessment of skin flakes

SUMMARY:
The principal objective of the study is the evaluation of the role of Human Papilloma Virus (HPV) in plantar warts (prevalence, genotype), resistant or not, treated or not, cured or not. This epidemiological study is an ancillary study of the prospective, randomized controlled, clinical study VRAIE (sponsor: APHP) comparing 5 usual strategies in the management of plantar warts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years or more.
* Clinical evaluation
* Number of warts lower than 10 on the 2 feet and total diameter of warts lower than 10 cm, whether previously treated or not
* In treated patients, all potentially active treatment on warts since at least one month should be stopped.
* Effective contraception for women of childbearing age
* Immunocompetent patients
* Patient with one or more warts on soles and board feet.

  * MYRMECIE : rounded warts, deep, covered with a stratum corneum more or less thick; after stripping, appear black points, very specific; often painful to pressure. They are lonely, single or not. They could regroup galley thick. The stripping can them to individualize.
  * Mosaic : plate small warts, superficial, often sitting on the heel or Forefoot. Little painful, they are often ignored by the patients when they appear
* Patient affiliated to the French social security.viral

Exclusion Criteria:

* Patient suspected to be immunocompromised
* Patient aged under 18 years
* Patient refusing to sign the consent
* Pregnant or lactating women
* Plantar calluses
* Known hypersensitivity to imiquimod (Aldara®) or any excipients of the cream (isostearic acid, benzyl alcohol, cetyl alcohol, stearyl alcohol, paraffin, polysorbate 60, sorbitan stearate, glycerol, methyl hydroxybenzoate, propyl hydroxybenzoate, xanthan gum, purified water)
* Known hypersensitivity to 5 fluoro-uracil (Efudix®) or any excipients of gel (stearyl alcohol, Vaseline, polysorbate 60, propyleneglycol, purified water - conservatives: METHYL PARAHYDROXYBENZOATE, PROPYL PARAHYDROXYBENZOATE)
* Contra-indication to Pomade M.O Cochon® (Known allergy to any components)
* Known hypersensitivity to Blenderm®
* Extra plantar concomitant warts (to exclude risk of endogenous recontamination by an extra plantar site)
* Plantar hyperhidrosis making impossible adhesion of plaster.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2000 skin flakes to be collected from patients included in VRAIE study
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Detection of HPV viral DNA on samples | up to Day 90
  research of positive HPV status

SECONDARY OUTCOMES:
Distribution of viral genotypes | up to Day 90
  number of samples containing one or more viral type (type 1, 2, 4 or mix)
Clinical remission defined | up to Day 90
  complete remission of wards confirmed by the physician, no later than day 90
Viral remission for patients with wards resistant to treatments | up to Day 90
  viral status modification from negative to positive between day 0 and day 30, day 60 or no more than day 90.
Clinical relapse | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: François Aubin, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon

IPD SHARING:
Plan to Share IPD: No